CLINICAL TRIAL: NCT02609334
Title: A Double-Blind, Randomised, Placebo-controlled, Cross-over, Phase 2 Mannitol Challenge Trial, Investigating the Efficacy of CRD007 in Adult Subjects With Asthma
Brief Title: RSPR-007 Mannitol Challenge Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RSPR Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RSPR-007
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo tables are given as a single dose
  Interventions: Other: Placebo
- CRD007 Low dose (Active Comparator): "Low dose" of CRD007 (pemirolast sodium) given as a single dose
  Interventions: Drug: CRD007
- CRD007 High dose (Active Comparator): "High dose" CRD007 (pemirolast sodium) given as a single dose
  Interventions: Drug: CRD007

INTERVENTIONS:
Drug: CRD007 — One single dose given 3 hours prior to Mannitol challenge
  Other Names: Pemirolast sodium
  Arms: CRD007 High dose; CRD007 Low dose
Other: Placebo — One single dose given 3 hours prior to Mannitol challenge
  Arms: Placebo

SUMMARY:
This is a double-blind, randomised, placebo-controlled, cross-over, Phase 2 trial evaluating two doses (a low and a high) of CRD007 for the treatment of asthmatic trial subjects with a positive asthma test (mannitol challenge) prior to enrolment.

DETAILED DESCRIPTION:
The present trial will include subjects with diagnosed asthma in a provocation model which mimics assessments of asthma control. Mannitol challenge is an indirect asthma provocation test, which requires the presence of inflammatory cells, particularly mast cells, in the airways.

The trial involved in total 5 subject visits and will last for a maximum of 30 days for each subject from Visit 2 (Randomisation) to Visit 5 (Follow up).

Visit 2,3, and 4 will be treatment visits where Investigational Medicinal Product (IMP) is administrated 3 hours before the Mannitol challenge.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 and <50 years
* Diagnosis of asthma

Exclusion Criteria:

* Clinical significant comorbidities
* Lower respiratory tract infection <6 weeks prior to Visit 1
* Others, as specified in the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
PD15 for mannitol after treatment with CRD007 and placebo | Forced expiratory volume at one second (FEV1) manoeuvres are performed 60 seconds after each dose
  The FEV1 value taken after the 0 mg capsule is taken as pre-challenge FEV1 and used to calculate the percentage decrease in FEV1 in response to the mannitol challenge. The test ends when the FEV1 has fallen by 15% or more (PD15)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, MD, Principal Investigator — Bispebjerg Hospital
Locations (2):
- Denmark (2):
  - Hvidovre Hospital, Hvidovre
  - Bisbebjerg Hospital, København NV